CLINICAL TRIAL: NCT00503282
Title: Urinary Catheter Exchange on Admission of Septic Elderly With Permanent Catheter Before Initiation of Antibiotics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: uc.ctil
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Fever; Heart Rate; Blood Pressure; C-Reactive Protein; Erythrocyte Sedimentation Rate
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the era of emerging antibiotics resistant microbiology, we look for better outcome in the treatment of infections in the elderly.

We look for guidelines to manage an elderly who has a permanent urinary catheter, admitting to E.R. with Fever/Sepsis.

We assume that exchanging the permanent urinary catheter prior to the Urine Culture sample as well as for initiating antibiotic treatment will improve the outcome of the patients.It could help the day-to-day fight for the proper antibiotics treatment to avoid resistance.

ELIGIBILITY:
Inclusion Criteria:

* >65 years
* Permanent Urinary Catheter
* FEVER or Septic State

Exclusion Criteria:

* Supra-Pubic Aspiration Catheters
* Septic Shock
* I.V. Antibiotics Initiated before admission

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2007-10; Study Completion 2007-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ben - Itzhak, Principal Investigator — HEBREW UNIVERSITY, JERUSALEM